CLINICAL TRIAL: NCT04765878
Title: RespirAq Humidification During Post-operative Invasive Mechanical Ventilation in Scheduled Cardiothoracic Surgical Patients: a Feasibility Study
Brief Title: RespirAq Humidifier Usability During Invasive Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Auckland University of Technology (Other)
Collaborators: Ministry of Business, Innovation and Employment (Unknown); Waikato District Health Board (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Humidification (Experimental)
  Interventions: Device: RespirAq Humidification

INTERVENTIONS:
Device: RespirAq Humidification — Humidifier

SUMMARY:
This study aims to capture preliminary safety and effectiveness information on a near-final humidifier device design and to provide data for more extensive research, if required. This feasibility study will investigate the following: process, resources, management, and scientific aspects of delivering humidification by the RespirAq humidifier device in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for coronary artery bypass surgery (CABG) will be recruited before their surgical procedure at the Waikato district health board during February, March, and April of 2021.

Exclusion Criteria:

* Age <18 years
* Have any other condition which, at the investigator's discretion, is believed may present a safety risk or impact the feasibility of the study or the study results
* Patients admitted for emergency CABG surgery
* Unable to provide written informed consent before surgery
* Patients who would be contra-indicated to HME humidification devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Temperature | max 24 hours
  Meet ISO standard
Humidity | max 24 hours
  Meet ISO standard

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Moylan, Principal Investigator — Auckland University of Technology